CLINICAL TRIAL: NCT02168296
Title: Exploratory Study to Assess the Pharmacokinetics in Relation to Blood Glucose and Insulin Levels After Intake of a Plant-based Ingredient in Healthy Subjects
Brief Title: Pharmacokinetics of Plant-based Ingredient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: FDS-NAA-1602
Record Dates: First submitted 2014-04-29; First posted 2014-06-20 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Blood glucose; subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- No added Plant-based ingredient (Placebo Comparator): No Plant-based ingredient added to starchy meal
  Interventions: Dietary Supplement: No Plant-based ingredient
- Low dose added to starchy meal (Active Comparator): Plant-based ingredient in low dose added to starchy meal
  Interventions: Dietary Supplement: Plant-based ingredient added to starchy meal
- High dose added to starchy meal (Active Comparator): Plant-based ingredient in high dose added to starchy meal
  Interventions: Dietary Supplement: Plant-based ingredient added to starchy meal
- Low dose added to liquid (Active Comparator): Plant-based ingredient in low dose added to liquid
  Interventions: Dietary Supplement: Plant-based ingredient added to liquid
- High dose added to liquid (Active Comparator): Plant-based ingredient in high dose added to liquid
  Interventions: Dietary Supplement: Plant-based ingredient added to liquid

INTERVENTIONS:
Dietary Supplement: Plant-based ingredient added to starchy meal
  Arms: High dose added to starchy meal; Low dose added to starchy meal
Dietary Supplement: Plant-based ingredient added to liquid
  Arms: High dose added to liquid; Low dose added to liquid
Dietary Supplement: No Plant-based ingredient
  Arms: No added Plant-based ingredient

SUMMARY:
The study is designed to explore the pharmacokinetics of a Plant-based ingredient in two different matrices, at different dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, age at start of the study 20 and 50 years
* Body mass index (BMI) ≥ 20,0 and ≤ 25,0 kg/m2
* Apparently healthy: no medical conditions which might affect the study measurements, absorption, metabolism and distribution (including diabetes type 1 and type 2, gastrointestinal dysfunction, gastrointestinal surgery and inflammatory diseases)
* Fasting blood glucose value of subjects is ≥ 3.4 and ≤ 6.1 mmol/litre (i.e. 62-110 mg/dl) at screening

Exclusion Criteria:

* Any history of diabetes, hyper- (or hypo-) glycemia or other disorder of glucose metabolism
* Any history of gastro-intestinal disorders (including frequent diarrhoea for example)
* Blood donation in the past 2 months
* Reported participation in another nutritional or biomedical trial 3 months before the pre-study examination or during the study
* Reported intense sporting activities > 10 h/w
* Consumption of > 21 alcoholic drinks in a typical week
* Not being used to eat breakfast
* Reported use of any nicotine containing products in the six months preceding the study and during the study itself
* Use of medication which interferes with study measurements
* Reported dietary habits: medically prescribed diet, slimming diet
* Not used to eat 3 meals a day
* Vegetarian
* Reported weight loss/gain (>10%) in the last six month before the study;
* Allergy or intolerance to food products and aversion to food products;

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
AUC of the plant based ingredient calculated by a non-compartmental model | predose, 15min, 30min, 45min, 1h, 1.5hrs, 2hrs, 3hrs, 5hrs, 8hrs, 12hrs.

SECONDARY OUTCOMES:
AUC of the plant based ingredient calculated by a compartmental model | predose, 15min, 30min, 45min, 1hr, 1.5hrs, 2hrs, 3hrs, 5hrs, 8hrs, 12hrs.
Urinary excretion of Plant-based ingredient | 24 hours

OTHER OUTCOMES:
AUC of the plant based ingredient calculated by a population model | predose, 15min, 30min, 45min, 1hr, 1.5hrs, 2hrs, 3hrs, 5hrs, 8hrs, 12hrs.
Describe the time course of the effect on glucose and insulin levels in response to the intake of plant based ingredient | predose, 15min, 30min, 45min, 1hr, 1.5hrs, 2hrs, 3hrs, 5hrs, 8hrs, 12hrs.
+iAUC Blood glucose | 120 minutes and 180 minutes
+iAUC Insulin | 120 minutes and 180 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins OPTIMED, Gierre, France